CLINICAL TRIAL: NCT00654329
Title: Dexmedetomidine for Peri-operative Sedation and Analgesia in Children Undergoing Bilateral Myringotomy With Tube Placement (BMT)
Brief Title: Dexmedetomidine vs Fentanyl for BMT
Acronym: DexBMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Julia C. Finkel, MD, Children's National Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3641; Agreement # 10698
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-03

CONDITIONS: Otitis
Keywords: Dexmedetomidine, transmucosal, myringotomy,
MeSH Terms: conditions — Otitis | interventions — Sodium Chloride; Saline Solution; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dexmedetomidine 1microgram/kilogram (Experimental): Dexmedetomidine 1microgram/kilogram intranasal
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 2 micrograms/kilogram (Experimental): Dexmedetomidine 2 micrograms/kilogram intranasal
  Interventions: Drug: Dexmedetomidine
- Fentanyl 2 micrograms/kilogram (Active Comparator): Fentanyl 2 micrograms/kilogram intranasal
  Interventions: Drug: Fentanyl
- Normal saline placebo (Placebo Comparator): Normal saline placebo intranasal
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — Normal saline, given intranasally
  Other Names: Normal Saline
  Arms: Normal saline placebo
Drug: Fentanyl — Fentanyl, nasal transmucosal, 2 micrograms/kilogram
  Other Names: Actiq, Fentora
  Arms: Fentanyl 2 micrograms/kilogram
Drug: Dexmedetomidine — Dexmedetomidine, transmucosal, 1 microgram/kilogram
  Other Names: Precedex
  Arms: Dexmedetomidine 1microgram/kilogram
Drug: Dexmedetomidine — Dexmedetomidine, 2 microgram/kilogram, transmucosal route
  Other Names: Precedex
  Arms: Dexmedetomidine 2 micrograms/kilogram

SUMMARY:
A randomized controlled clinical trial to examine effects of intranasal dexmedetomidine, an α2-adrenorecptor agonist, on pain control and agitation in children undergoing BMT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation:

  1. The subject is 6 months to 6 years of age
  2. The subject's American Society of Anesthesiologists (ASA) physical status is ASA 1 or 2 (see appendix 1)
  3. The subject is scheduled for elective bilateral myringotomy with tube placement
  4. The subject's parent/legally authorized guardian has given written informed consent to participate

     Exclusion Criteria:
* Subjects will be excluded from study participation if any of the following exclusion criteria exists:

  1. The subject has a history or a family (parent or sibling) history of malignant hyperthermia
  2. The subject has known significant renal or hepatic disorders determined by medical history, physical examination or laboratory tests
  3. The subject has a known or suspected allergy to opioid analgesics or dexmedetomidine
  4. The subject has history of. cardiovascular issues which would preclude the use of dexmedetomidine, (e.g. Down's Syndrome, dysrhythmias, conditions where hypotension is to be avoided)
  5. The subject has know central nervous system disease or neurological impairment
  6. The subject is an ASA classification of 3 or greater (See Appendix 1)
  7. The subject has a medical condition requiring an intravenous induction (i.e. severe uncontrolled gastro-esophageal reflux)
  8. The subject refuses inhalation induction
  9. The subject is scheduled for a surgical sub-procedure (i.e. adenoidectomy, tonsillectomy)

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine 1microgram/Kilogram: Dexmedetomidine 1microgram/kilogram (mcg/kg) intranasal
- Dexmedetomidine 2 Micrograms/Kilogram: Dexmedetomidine 2 micrograms/kilogram (mcg/kg) intranasal
- Fentanyl 2 Micrograms/Kilogram: Fentanyl 2 micrograms/kilogram (mcg/kg) intranasal
Period: Overall Study
Arm/Group | Dexmedetomidine 1microgram/Kilogram | Dexmedetomidine 2 Micrograms/Kilogram | Fentanyl 2 Micrograms/Kilogram | Normal Saline Placebo
Started | 23 | 28 | 23 | 27
Completed | 23 | 28 | 23 | 27
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine 1microgram/Kilogram | Dexmedetomidine 2 Micrograms/Kilogram | Fentanyl 2 Micrograms/Kilogram | Normal Saline Placebo | Total
Number analyzed (Participants) | 23 | 28 | 23 | 27 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 28 | 23 | 27 | 101
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 1.92 (.94) | 2.17 (1.51) | 2.25 (1.47) | 2.17 (1.66) | 2.14 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 10 | 10 | 35
  Male | 18 | 18 | 13 | 17 | 66
Region of Enrollment [Number; unit: participants]
  United States | 23 | 28 | 23 | 27 | 101

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pain
Description: Pain greater than a zero reported in the Post Anesthesia Care Unit (PACU)
Time Frame: up to 24 hours
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine 1microgram/Kilogram | Dexmedetomidine 2 Micrograms/Kilogram | Fentanyl 2 Micrograms/Kilogram | Normal Saline Placebo
Number analyzed (Participants) | 23 | 28 | 23 | 27
participants | 6 | 11 | 7 | 18

2. Secondary Outcome: Length of Stay in PACU
Description: Total time from PACU entry until discharge
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine 1microgram/Kilogram | Dexmedetomidine 2 Micrograms/Kilogram | Fentanyl 2 Micrograms/Kilogram | Normal Saline Placebo
Number analyzed (Participants) | 23 | 28 | 23 | 27
minutes | 48 (26) | 88 (69) | 46 (25) | 48 (27)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine 1microgram/Kilogram | Dexmedetomidine 2 Micrograms/Kilogram | Fentanyl 2 Micrograms/Kilogram | Normal Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/28 | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 0/23 | 1/28 | 0/23 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dexmedetomidine 1microgram/Kilogram (N=23) | Dexmedetomidine 2 Micrograms/Kilogram (N=28) | Fentanyl 2 Micrograms/Kilogram (N=23) | Normal Saline Placebo (N=27)
Bradycardia (Cardiac disorders) | 0/0 (0) | 1/1 (1) | 0/0 (0) | 0/0 (0) — Heart rate dropped to 42 bpm for 2 min post-op.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes